CLINICAL TRIAL: NCT01303094
Title: Phase II Randomized Trial to Evaluate Two Strategies: Continuing Versus Intermittent (Drug-holiday) Trabectedin-regimen in Patients With Advanced Soft Tissue Sarcoma Experiencing Response or Stable Disease After the Sixth Cycle
Brief Title: Continuing vs Intermittent Trabectedin in Patients With Advanced Soft Tissue Sarcoma
Acronym: T-DIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Collaborators: French Sarcoma Group (Other); Study Group of Bone Tumors (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T-DIS-1001
Record Dates: First submitted 2011-02-23; First posted 2011-02-24 (Estimated); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Soft Tissue Sarcoma; Uterine Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Trabectedin; Treatment Interruption

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuation of Trabectedin (Other): patient receives 6 cycles of trabectedin, then one dose 15 days after the 6th cycle, every 3 weeks until progression/ toxicity
  Interventions: Drug: Trabectedin
- "Drug holiday" therapy (Other): patient receives 6 cycles of trabectedin, then one dose 15 days after the 6th cycle and he stops the drug until progression and re-challenge
  Interventions: Other: Drug: holiday

INTERVENTIONS:
Drug: Trabectedin — Trabectedin will be administered without drug holiday in Arm A until unacceptable toxicity, progressive disease or patient decision. The treatment beyond disease progression and in case of intolerance will be decided according to investigator discretion. In case of progression after drug discontinuation by patient decision, a re-challenge of Trabectedin is possible.
  Other Names: Yondelis
  Arms: Continuation of Trabectedin
Other: Drug: holiday — A drug-holiday will start after the 6th cycle until disease progression, and then Trabectedin will be re-challenged. Trabectedin will be administered until unacceptable toxicity, second evidence of progressive disease or patient decision.
  Other Names: No drug
  Arms: "Drug holiday" therapy

SUMMARY:
This randomization discontinuation trial will allow for concomitant evaluation of the following:

* Side effects and benefits of immediate continuation of Trabectedin after the sixth cycle
* Side effects and benefits of a drug holiday

DETAILED DESCRIPTION:
Selection part (220 patients):

Trabectedin (depending on dose reductions : between 1.5 and 1 mg/m²/3 weeks; over 24 hour administration) until progression, intolerance or 6 cycles (according to the SPC of Trabectedin)

Randomized part (50 patients):

After the 6 first cycles, if there is not progression or unacceptable toxicity, the patients will be randomly assigned to continuous or "intermittent/holiday" therapy with CT-scan evaluation every 6 weeks in both arms

* Arm A Continuation of Trabectedin (between 1.5 and 1 mg/m²/3 weeks; over 24 hour administration) until progression or intolerance
* Arm B "Intermittent/holiday" therapy. Rechallenge of Trabectedin will be implemented in the event of progression; in this case administration of Trabectedin will occur until the second progression or intolerance

ELIGIBILITY:
Inclusion Criteria (for the selection part):

* Inoperable or metastatic soft tissue sarcoma and/or uterine sarcoma
* Measurable lesions (RECIST 1.1)
* Performance status ≤ 2
* Age ≥ 18
* Normal hematological parameters (polynuclear neutrophils ≥ 1500, hemoglobin level ≥ 9 g/dl, platelets counts ≥ 100,000)
* Adequate biological parameters :
* Adequate hepatic function (bilirubin ≤ ULN , SGPT/ALT and SGOT/AST ≤ 2.5 x ULN)
* Alkaline phosphatases ≤ 2.5 x ULN, If Alkaline phosphatases ≥ 2.5 ULN, hepatic isoenzymes 5-nucleotidases or GGT tests must be performed; hepatic isoenzymes 5- nucleotidases and/or GGT must be within the normal range
* Albumin ≥ 25 g/L
* Adequate renal function : Serum creatinine ≤ 1.5 x ULN
* Creatine phosphokinase ≤ 2.5 x ULN
* Adequate central venous access
* Pregnant or lactating women or men of reproductive potential must use effective contraceptive methods
* Patient covered by government health insurance
* Information sheet given to the patient (Patient information sheet 1)

Exclusion Criteria (for the selection part):

* Patients that have received more than one regimen of chemotherapy for metastatic or inoperable soft tissue or uterine sarcoma, after the failure/intolerance of doxorubicin and ifosfamide. Maintenance treatment does not count as treatment line
* The following histological subtypes : GIST, rhabdomyosarcoma, aggressive fibromatosis, desmoïd tumour, PNET, carcinosarcoma, and all bone sarcomas
* Single tumour in an irradiated region
* Other malignant tumour over the past five years (except basal cell carcinoma or cervical carcinoma in situ adequately treated)
* Currently active bacterial or fungus infection (> grade 2 CTC [CTCAE] Version 4.02). Known HIV1, HIV2, hepatitis B or hepatitis C infections
* Presence of known leptomeningeal or brain metastasis
* Patients unable to receive corticotherapy
* Any circumstance that could jeopardise compliance or proper follow-up during the trial
* Pregnant or nursing women

Inclusion Criteria (for the randomized part):

* Patient registered in the selection part
* Stable tumour or objective response (CR + PR) after 6 Trabectedin (Yondelis®) cycles, according to local assessment
* Available copies of thoraco-abdominal and pelvic scan performed prior to the first cycle and after the sixth cycle
* Performance status ≤ 2
* Patients receiving at least 1 mg/m²/3 weeks of Trabectedin at the time of the sixth cycle
* Normal hematological parameters (polynuclear neutrophils ≥ 1500, hemoglobin level ≥ 9 g/dl, platelets counts ≥ 100,000)
* Adequate biological parameters :
* Adequate hepatic function (bilirubin ≤ ULN , SGPT/ALT and SGOT/AST ≤ 2.5 x ULN)
* Alkaline phosphatases ≤ 2.5 x ULN, If Alkaline phosphatases ≥ 2.5 ULN, hepatic isoenzymes 5-nucleotidases or GGT tests must be performed; hepatic isoenzymes 5- nucleotidases and/or GGT must be within the normal range
* Albumin ≥ 25 g/L
* Adequate renal function : Serum creatinine ≤ 1.5 x ULN
* Creatine phosphokinase (CPK) ≤ 2.5 x ULN
* Adequate central venous access
* Pregnant or lactating women or men of reproductive potential must use effective contraceptive methods
* Informed consent form signed by the patient or the patient's legal representative (patient information sheet 2 and informed consent)

Exclusion Criteria (for the randomized part):

* Tumour progression (according to RECIST 1.1) during the first six Yondelis cycles
* Non-availability of baseline scans prior to the first cycle and following the sixth cycle
* Currently active bacterial or fungus infection (> grade 2 CTC [CTCAE] Version 4.02). Known HIV1, HIV2, hepatitis B or hepatitis C infections
* Presence of known leptomeningeal or brain metastasis
* Creatinine clearance less than 30 ml/min
* Patients unable to receive corticotherapy
* Any circumstance that could jeopardise compliance or proper follow-up during the trial
* Pregnant or nursing women
* Hypersensitivity to Trabectedin or any excipient in prior cycles

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2018-08-09 (Actual)

PRIMARY OUTCOMES:
PFS rate 24 weeks after randomization | 24 weeks after randomization
  In each arms among non progressive patients after the 6 first cycles of Trabectedin : occurrence of progression or death 24 weeks after the date of randomization. Intention to treat analysis. Centralised radiological review.

SECONDARY OUTCOMES:
Response rate | 6, 12 and 18 weeks after randomization
  stabilisation, complete and partial responses according to RECIST 1.1
Progression free survival rates | 12 and 54 weeks after randomization
  According to RECIST 1.1
Survival rates | 12 and 24 months after randomization
Median progression-free and median overall survivals | Up to 5 years after randomization
Tolerability - safety | Up to 30 days after the last study drg administration
  According to NCI-CTC V4.0 scale
Clinical and biological predictive factors for non progression at the 6th cycle | At baseline
  Collected data at baseline : age, gender, comorbidity, disease history, previous treatment, tumor description, biological parameters
Post-randomization cost of care | For one year after randomization
  Cost of care will be evaluated by macro-costing approach
Self estimation of general health status | For 1 year after randomization
  Evaluation every 6 weeks by 100-mm-long horizontal visual analog scale (VAS) that ranged from worst imaginable health (as bad as death, 0) to perfect health

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas PENEL, MD, PhD, Principal Investigator — Centre Oscar Lambret
Locations (16):
- France (16):
  - Saint-Jacques Hospital, Besançon
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Léon Bérard Center, Lyon
  - Centre Léon Bérard, Lyon
  - Paoli Calmette Institute, Marseille
  - CHU Timone Adultes, Marseille
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - Centre Henri Becquerel, Rouen
  - Centre René Huguenin, Saint-Cloud
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Le Cesne A, Blay JY, Domont J, Tresch-Bruneel E, Chevreau C, Bertucci F, Delcambre C, Saada-Bouzid E, Piperno-Neumann S, Bay JO, Mir O, Ray-Coquard I, Ryckewaert T, Valentin T, Isambert N, Italiano A, Clisant S, Penel N. Interruption versus continuation of trabectedin in patients with soft-tissue sarcoma (T-DIS): a randomised phase 2 trial. Lancet Oncol. 2015 Mar;16(3):312-9. doi: 10.1016/S1470-2045(15)70031-8. Epub 2015 Feb 11. PMID 25680558